CLINICAL TRIAL: NCT00568464
Title: Phase II Study of VCD/IE in the Treatment of the Patients With Ewing's Sarcoma Family of Tumors
Brief Title: Study on VCD/IE in the Patients With Ewing's Sarcoma Family of Tumors (ESFT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrollment is slower than expected
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCD/IE-ESFT
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Ewing's Sarcoma
Keywords: ESFT (Ewing's sarcoma family of tumors); Response rate; TTP; OS; Toxicity
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: VCR, CTX, ADM; IFO, VP-16

INTERVENTIONS:
Drug: VCR, CTX, ADM; IFO, VP-16 — VCD: VCR 2 mg d1, CTX 1200 mg/m2 d1, Mesna 240 mg/m2 tid d1, ADM 75mg/m2 d1, G-CSF 300 ug/d d5-11; IE: IFO 1800mg/m2 d1-5,Mesna 360 mg/m2 tid d1-5,VP-16 100 mg/m2 d1-5,G-CSF 300 ug/d d6-12; q3w. Surgery or radiation will be done to the patients with local diseases after four cycles of VCD/IE.
  Other Names: VCD/IE

SUMMARY:
The purpose of this clinical trial was to evaluate the efficacy and tolerability of the sequential therapy of VCD/IE in the patients with ESFT.

DETAILED DESCRIPTION:
80-90% patients of ESFT will develope disease progression during the period of local treatment (surgery or radiation). The survival has been improved in these 30 years due to chemotherapy. VCD/IE is widely used in the world for the patients with ESFT, but it is rarely used in China due to its high dosage.

ELIGIBILITY:
Inclusion Criteria:

* Age range 10-65 years old
* Histological confirmed ESFT
* No previous therapy
* ECOG performance status less than 2
* Life expectancy of more than 12 weeks
* Normal laboratory values: hemoglobin>8.0g/dl, neutrophil>2×109/L, platelet > 80×109/L, Hb > 80×1012/L, serum creatine < 1×upper limitation of normal(ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN

Exclusion Criteria:

* Pregnant or lactating women
* Received treatment for the disease previously
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis and bone marrow involvement
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* History of allergy to the drugs in this trial
* Abnormal LVEF level

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Response Rate | every two cycles

SECONDARY OUTCOMES:
Toxicity | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China